CLINICAL TRIAL: NCT03441022
Title: Continuous Data Collection and Analysis for Stroke Prevention Using a Wearable Sensor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain equipment from Sponsor to be able to proceed with the study.
Sponsor: Mayo Clinic (Other)
Collaborators: Koronis Biomedical Technologies (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Suraj Kapa, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-006346; 1R43AG058516-01 (NIH)
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
Keywords: Cardioversion; BodyGuardian; Amiigo Wristband
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electric Countershock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cardioversion (Experimental): Amiigo watch during atrial fibrillation cardioversion. Optional sub-study: additional 30 days wearing Amiigo watch as well as BodyGuardian device.
  Interventions: Device: Amiigo Watch Only; Device: Amiigo Watch + BodyGuardian

INTERVENTIONS:
Device: Amiigo Watch Only — Subjects will be asked to wear a wrist band with capabilities to detect their heart rate or rhythm on the basis of PPG on either wrist around the time of their cardioversion procedure. Data will be acquired from the wrist band at the same time as the electrocardiogram (ECG) monitor to which subjects are hooked up for the purposes of the cardioversion.
  Other Names: Cardioversion
Device: Amiigo Watch + BodyGuardian — Subjects will be sent home after the cardioversion with a 30 day heart monitor called the BodyGuardian. This device continuously monitors their heart rate and rhythm and they will wear this on the chest. Subjects will also wear the wrist monitor over the same 30 day period.
  Other Names: Cardioversion plus 30 days

SUMMARY:
The purpose of this study is to determine whether a wristband that detects your pulse can detect your heart rate and rhythm similar to electrocardiograms (ECG).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a wristband that detects your pulse can detect your heart rate and rhythm similar to electrocardiograms (ECG). These wristbands detect your pulse based on a technique called "photoplethysmography," (PPG). PPG is a common method in which an individual's pulse is detected based on a light signature interpreted by the wristband. Most commercially available heart rate monitors use PPG to determine your heart rate, but the accuracy is variable.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older with a primary diagnosis of atrial fibrillation
2. Willing and able to provide informed consent and follow the study protocol
3. Clinically indicated planned restoration of normal rhythm

Exclusion Criteria:

1. Unable to provide informed consent
2. Unable to follow the study protocol
3. Women who are pregnant
4. Subjects with implantable devices (only if participating in phase 2-BodyGuardian processes/testing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Watch Accuracy during Cardioversion | Duration of cardioversion procedure
  Determine whether the R-R interval estimate from artifact-free non-invasive photoplethysmography sample waveform segments is a reasonable basis for a atrial fibrillation (AF) detection algorithm as compared to a gold standard measurement from ECG in the acute cardioversion setting
Watch Accuracy compared to BodyGuardian | 30 days
  Determine the accuracy of ambulatory photoplethysmography for detection of heart rhythm when compared with a wearable clinically available 30 day monitor (BodyGuardian) in terms of accuracy of AF detection.

CONTACTS AND LOCATIONS:
Overall Officials: Suraj Kapa, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials